CLINICAL TRIAL: NCT00081263
Title: A Randomized Double-Blind Phase II Trial of Celecoxib, A COX-2 Inhibitor, in the Treatment of Patients With Cervical Intraepithelial Neoplasia 2/3 or 3 (CIN 2/3 or 3)
Brief Title: Celecoxib in Treating Patients With Cervical Intraepithelial Neoplasia
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Gynecologic Oncology Group (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Organization: GOG Foundation (Network)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: GOG-0207; NCI-2009-00583 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); CDR0000360805; GOG-0207 (Other: NRG Oncology); GOG-0207 (Other: DCP); GOG-0207 (Other: CTEP); U10CA101165 (NIH)
Record Dates: First submitted 2004-04-07; First posted 2004-04-08 (Estimated); Results first posted 2017-09-15 (Actual); Last update posted 2017-09-15 (Actual); Status verified 2017-08

CONDITIONS: Cervical Carcinoma; Cervical Intraepithelial Neoplasia Grade 2/3; Stage 0 Cervical Cancer
MeSH Terms: conditions — Uterine Cervical Neoplasms; Uterine Cervical Dysplasia | interventions — Celecoxib

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Arm I (celecoxib) (Experimental): Patients receive oral celecoxib once daily for 14-18 weeks.
  Interventions: Drug: Celecoxib; Other: Laboratory Biomarker Analysis
- Arm II (placebo) (Placebo Comparator): Patients receive oral placebo once daily for 14-18 weeks.
  Interventions: Other: Laboratory Biomarker Analysis; Other: Placebo

INTERVENTIONS:
Drug: Celecoxib — Given orally
  Other Names: Benzenesulfonamide, 4-[5-(4-methylphenyl)-3-(trifluoromethyl)-1H-pyrazol-1-yl]-; Celebrex; SC-58635; YM 177
  Arms: Arm I (celecoxib)
Other: Laboratory Biomarker Analysis — Correlative studies
Other: Placebo — Given orally
  Other Names: placebo therapy; PLCB; sham therapy
  Arms: Arm II (placebo)

SUMMARY:
This randomized phase II trial studies how well celecoxib works in treating patients with cervical intraepithelial neoplasia, a precancerous lesion of the cervix which can develop into cervical cancer. Celecoxib may be effective in preventing the development of cervical cancer in patients who have cervical intraepithelial neoplasia.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine the efficacy of celecoxib to induce complete remission (or partial regression to cervical intraepithelial neoplasia (CIN) 1) of CIN 2/3 or CIN 3 as evaluated in the post-treatment excisional biopsy.

II. To determine the toxicity of celecoxib (400 mg once daily) as assessed by Common Terminology Criteria for Adverse Events in this patient population of women with CIN 2/3 or CIN 3.

SECONDARY OBJECTIVES:

I. To assess whether treatment with celecoxib changes the number of quadrants containing acetowhite lesions as determined through colposcopic examination.

II. To determine the efficacy of celecoxib treatment in changing human papillomavirus (HPV) viral load in cervical cells.

III. To examine the association of histologic response; HPV viral load; lesion size; proliferation index (marker of proliferation Ki-67 [Ki67]), apoptosis index (terminal deoxynucleotidyl transferase (TdT)-mediated dUTP nick end labelin [TUNEL] assay), angiogenesis (vascular endothelial growth factor [VEGF]), and cyclooxygenase-2 (COX-2) in tissue; the amount of VEGF and basic fibroblast growth factor (bFGF) in serum before and after treatment; and the amount of celecoxib present in serum during treatment. Cervical cytology karyometry will be assessed as a potential marker for regression IV. To determine the feasibility of digital imaging, web-based review of histopathology in a Gynecologic Oncology Group (GOG) study.

V. To compare the diagnoses of the web-based review of histopathology with the diagnoses of GOG's standard procedure.

OUTLINE: Patients are randomized to 1 of 2 treatment arms.

ARM I: Patients receive oral celecoxib once daily for 14-18 weeks.

ARM II: Patients receive oral placebo once daily for 14-18 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have histologically proven CIN 2/3 or CIN 3 diagnosed by cervical biopsy between 2 and 8 weeks prior to enrollment

  * For a patient to be eligible, the pathology report must clearly state "CIN 2/3" or "CIN 3" or must state "moderate-severe dysplasia", "moderate-severe dyskaryosis," "severe dysplasia," or "severe dyskaryosis;" patients with a diagnosis of CIN 2 alone or moderate dysplasia or dyskaryosis alone are not eligible for this study (3/26/2007)
* Patients must have a satisfactory (readable, good quality) colposcopic evaluation at least 14 days after diagnostic biopsy
* Patients must have signed an approved informed consent and authorization permitting release of personal health information
* Patients must have colposcopically visible cervical lesion at entry consistent with biopsy
* Patients must have a negative urine pregnancy test; women of childbearing potential must practice an acceptable form of contraception (e.g. intrauterine device, contraceptive pills, diaphragm, condoms)
* Patients must have a GOG Performance Status of 0, 1, or 2
* Patients must agree to refrain from using non-steroidal anti-inflammatory drugs (NSAIDS) and aspirin during the time they are taking the study medication
* Patients must be good candidates for delayed treatment of their CIN, i.e. they must be reliable to return for follow-up and provide a combination of at least three phone numbers or addresses for contact
* Hemoglobin (HgB) greater than 11.0g/dl
* White blood cell (WBC) count greater than 3000/mcl
* Platelet count greater than 125,000/mcl (3/26/2007)
* Creatinine less than or equal to 1.5 x upper limit normal (ULN)
* Total bilirubin less than or equal to 1.5 x ULN excluding Gilbert's disease
* Aspartate aminotransferase (AST) and alanine aminotransferase (ALT) < 2.0 x ULN

Exclusion Criteria:

* Patients who are pregnant or lactating
* Patients with cytologic or biopsy evidence of endocervical dysplasia or invasive cancer
* Patients with undiagnosed abnormal vaginal bleeding
* Patients who have previously taken celecoxib or any other COX-2 inhibitor at a frequency of greater than 3 times per week within 2 months (60 days) prior to randomization; patients can use Naproxen without restriction (6/23/2008)
* Patients with a known immunocompromised condition
* Patients who have had a known allergic reaction to any NSAIDS or aspirin (asthma, urticaria, allergic-type reaction)
* Patients with a prior history of cervical cancer
* Patients with hypersensitivity to Celecoxib
* Patients with a known allergic reaction to sulfonamides
* Patients with a history of peptic ulcer disease
* Patients currently using fluconazole or lithium
* Patients with a chronic or acute renal, or hepatic disorder, a significant bleeding disorder, or any other condition which in the investigator's opinion might preclude study participation for the duration of the trial
* Patients with a history of transient ischemic attack (TIA), stroke, cardiovascular disease or uncontrolled hypertension

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 130 (Actual)
Dates: Start 2005-06; Primary Completion 2012-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Janet Rader, Principal Investigator — NRG Oncology
Locations (43):
- United States (43):
  - University of Arizona Cancer Center-North Campus, Tucson, Arizona
  - University of Arkansas for Medical Sciences, Little Rock, Arkansas
  - Beebe Medical Center, Lewes, Delaware
  - Christiana Care Health System-Christiana Hospital, Newark, Delaware
  - Carle Clinic-Urbana Main, Urbana, Illinois
  - Elkhart Clinic, Elkhart, Indiana
  - Michiana Hematology Oncology PC-Elkhart, Elkhart, Indiana
  - Elkhart General Hospital, Elkhart, Indiana
  - Community Howard Regional Health, Kokomo, Indiana
  - IU Health La Porte Hospital, La Porte, Indiana
  - Michiana Hematology Oncology PC-Mishawaka, Mishawaka, Indiana
  - Saint Joseph Regional Medical Center-Mishawaka, Mishawaka, Indiana
  - Michiana Hematology Oncology PC-Plymouth, Plymouth, Indiana
  - Memorial Hospital of South Bend, South Bend, Indiana
  - Michiana Hematology Oncology PC-South Bend, South Bend, Indiana
  - Northern Indiana Cancer Research Consortium, South Bend, Indiana
  - Michiana Hematology Oncology PC-Westville, Westville, Indiana
  - Union Hospital of Cecil County, Elkton, Maryland
  - Borgess Medical Center, Kalamazoo, Michigan
  - Bronson Methodist Hospital, Kalamazoo, Michigan
  - West Michigan Cancer Center, Kalamazoo, Michigan
  - Lakeland Hospital, Saint Joseph, Michigan
  - Marie Yeager Cancer Center, Saint Joseph, Michigan
  - University of Missouri - Ellis Fischel, Columbia, Missouri
  - Saint Louis University Hospital, St Louis, Missouri
  - Women's Cancer Center of Nevada, Las Vegas, Nevada
  - Rutgers New Jersey Medical School, Newark, New Jersey
  - Montefiore Medical Center - Moses Campus, The Bronx, New York
  - UNC Lineberger Comprehensive Cancer Center, Chapel Hill, North Carolina
  - Gynecologic Oncology Network, Greenville, North Carolina
  - FirstHealth of the Carolinas-Moore Regional Hosiptal, Pinehurst, North Carolina
  - Wake Forest University Health Sciences, Winston-Salem, North Carolina
  - University of Cincinnati, Cincinnati, Ohio
  - Case Western Reserve University, Cleveland, Ohio
  - Hillcrest Hospital Cancer Center, Mayfield Heights, Ohio
  - Lake University Ireland Cancer Center, Mentor, Ohio
  - University of Oklahoma Health Sciences Center, Oklahoma City, Oklahoma
  - Oklahoma Cancer Specialists and Research Institute-Tulsa, Tulsa, Oklahoma
  - Sanford USD Medical Center - Sioux Falls, Sioux Falls, South Dakota
  - Vanderbilt University/Ingram Cancer Center, Nashville, Tennessee
  - Brooke Army Medical Center, Fort Sam Houston, Texas
  - Carilion Clinic Gynecological Oncology, Roanoke, Virginia
  - Froedtert and the Medical College of Wisconsin, Milwaukee, Wisconsin

REFERENCES:
- [Derived] Rader JS, Sill MW, Beumer JH, Lankes HA, Benbrook DM, Garcia F, Trimble C, Tate Thigpen J, Lieberman R, Zuna RE, Leath CA 3rd, Spirtos NM, Byron J, Thaker PH, Lele S, Alberts D. A stratified randomized double-blind phase II trial of celecoxib for treating patients with cervical intraepithelial neoplasia: The potential predictive value of VEGF serum levels: An NRG Oncology/Gynecologic Oncology Group study. Gynecol Oncol. 2017 May;145(2):291-297. doi: 10.1016/j.ygyno.2017.02.040. Epub 2017 Mar 10. PMID 28285845

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Arm I (Celecoxib) | Arm II (Placebo)
Started | 67 | 63
Completed | 50 | 41
Not Completed | 17 | 22
Not completed — clerical error | 1 | 0
Not completed — wrong cell type | 7 | 5
Not completed — improper pre-protocol therapy | 0 | 1
Not completed — Inadequate pathology | 0 | 1
Not completed — Never treated | 4 | 5
Not completed — Inadequate data | 5 | 10

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm I (Celecoxib) | Arm II (Placebo) | Total
Number analyzed (Participants) | 50 | 41 | 91
Age, Customized [Count of Participants; unit: Participants]
  18-19 years | 1 | 5 | 6
  20-29 years | 30 | 23 | 53
  30-39 years | 13 | 10 | 23
  40-49 years | 6 | 3 | 9
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 50 | 41 | 91
  Male | 0 | 0 | 0
Cell Type [Count of Participants; unit: Participants] — Cell Type Definitions:
  Cervical Intraepithelial Neoplasia 2/3 is defined as moderate-severe dysplasia or moderate-severe dyskaryosis.
  Cervical Intraepithelial Neoplasia 3 is defined as severe dysplasia or severe dyskaryosis.
  Participants
    Cervical Intraepithelial Neoplasia 2/3 | 14 | 11 | 25
    Cervical Intraepithelial Neoplasia 3 | 36 | 30 | 66

OUTCOME MEASURES:

1. Primary Outcome: Histologic Regression
Description: Whether or not patients with CIN 2/3 or CIN 3 upon entry experience a complete remission (or partial regression to CIN 1) in the post-treatment excisional biopsy.
Time Frame: Post treatment evaluation was done 14 to 18 weeks after treatment randomization
Population: Eligible, Treated, and Evaluable patients
Measure: Number (90% Confidence Interval); unit: percentage of participants
Arm/Group | Arm I (Celecoxib) | Arm II (Placebo)
Number analyzed (Participants) | 50 | 41
percentage of participants | 40 [28 to 53] | 34.1 [22 to 48]

2. Primary Outcome: Incidence of Adverse Effects (Grade 3 or Higher) as Assessed by Common Terminology Criteria for Adverse Events Version 3.0
Description: Number of participants with a grade of 3 or higher during the treatment period.
Time Frame: Assessed every cycle while on treatment, 30 days after the last cycle of treatment
Population: Eligible and treated patients.
Measure: Number; unit: participants
Arm/Group | Arm I (Celecoxib) | Arm II (Placebo)
Number analyzed (Participants) | 50 | 41
participants
  Gastrointestinal | 1 | 0
  Pain | 0 | 1

3. Other Pre Specified Outcome: To Examine the Association of Histologic Response in COX-2 in Tissue
Time Frame: Up to 18 weeks
Reporting Status: Not Posted

4. Other Pre Specified Outcome: To Examine the Association of Histologic Response in HPV Viral Load in Serum Before and After Treatment
Time Frame: Up to 18 weeks
Reporting Status: Not Posted

5. Other Pre Specified Outcome: HPV Viral Load Before and After Treatment
Time Frame: Up to 18 weeks
Reporting Status: Not Posted

6. Other Pre Specified Outcome: To Examine the Association of Histologic Response in the Levels of Celecoxib in Serum During Treatment.
Time Frame: Up to 18 weeks
Reporting Status: Not Posted

7. Other Pre Specified Outcome: Levels of Serum bFGF
Time Frame: Up to 18 weeks
Reporting Status: Not Posted

8. Other Pre Specified Outcome: Levels of Serum VEGF
Time Frame: Up to 18 weeks
Reporting Status: Not Posted

9. Other Pre Specified Outcome: To Determine the Feasibility of Digital Imaging Using Pathologist's Diagnosis and Diagnostic Technique (Web-based or Standard Method).
Time Frame: Baseline
Reporting Status: Not Posted

10. Other Pre Specified Outcome: To Examine the Association of Histologic Response in Proliferation Index (Ki67).
Time Frame: Up to 18 weeks
Reporting Status: Not Posted

11. Other Pre Specified Outcome: Proportion of Patients Whose Eligibility Can be Successfully Determined Using the Web-based Review
Time Frame: Baseline
Reporting Status: Not Posted

12. Other Pre Specified Outcome: The Number of Quadrants Involving CIN
Time Frame: Up to 18 weeks
Reporting Status: Not Posted

13. Other Pre Specified Outcome: To Examine the Association of Histologic Response in Apoptosis Index (TUNEL Assay)
Time Frame: Up to 18 weeks
Reporting Status: Not Posted, anticipated posting 2099-01

14. Other Pre Specified Outcome: To Examine the Association of Histologic Response in Angiogenisis (VEGF)
Time Frame: Up to 18 weeks
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: All Adverse Events (AEs) occurring during treatment and up to 30 days after stopping the study treatment are reported.
Arm/Group | Arm I (Celecoxib) | Arm II (Placebo)
Serious Adverse Events (participants affected / at risk) | 0/67 | 1/63
Other Adverse Events (participants affected / at risk) | 25/67 | 25/63
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm I (Celecoxib) (N=67) | Arm II (Placebo) (N=63)
Inf W/Nml Or Gr 1 Or 2 ANC: Cervix (Infections and infestations) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Arm I (Celecoxib) (N=67) | Arm II (Placebo) (N=63)
Hemoglobin (Blood and lymphatic system disorders) | 1 | 0
Constitutional Symptoms - Other (General disorders) | 0 | 1
Sweating (General disorders) | 0 | 1
Weight Gain (General disorders) | 1 | 1
Fatigue (General disorders) | 1 | 2
Insomnia (General disorders) | 0 | 1
Rash (Skin and subcutaneous tissue disorders) | 0 | 1
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 1
Flatulence (Gastrointestinal disorders) | 2 | 2
Heartburn (Gastrointestinal disorders) | 5 | 3
Ulcer,gi - Stomach (Gastrointestinal disorders) | 1 | 0
Vomiting (Gastrointestinal disorders) | 1 | 2
Constipation (Gastrointestinal disorders) | 0 | 1
Nausea (Gastrointestinal disorders) | 3 | 6
Gastrointestinal - Other (Gastrointestinal disorders) | 0 | 1
Diarrhea (Gastrointestinal disorders) | 1 | 4
Hemorrhage, Gu - Vagina (Vascular disorders) | 1 | 2
Inf W/Nml Or Gr 1 Or 2 Anc: Upper Airway Nos (Infections and infestations) | 1 | 0
Inf Unknown Anc: Sinus (Infections and infestations) | 0 | 1
Edema: Limb (Blood and lymphatic system disorders) | 1 | 0
Dermal Change (Blood and lymphatic system disorders) | 2 | 3
Involuntary Movement (Nervous system disorders) | 0 | 1
Somnolence (Nervous system disorders) | 0 | 1
Dizziness (Nervous system disorders) | 0 | 3
Flashing Lights/Floaters (Eye disorders) | 0 | 1
Blurred Vision (Eye disorders) | 1 | 0
Pain - Other (General disorders) | 1 | 0
Pain: Throat/Pharynx/Larynx (General disorders) | 1 | 0
Pain: Head/Headache (General disorders) | 6 | 10
Pain: Stomach (General disorders) | 0 | 1
Pain: Abdominal Pain Nos (General disorders) | 4 | 7
Pain: Muscle (General disorders) | 0 | 1
Incontinence, Urinary (Renal and urinary disorders) | 0 | 1
Vaginal Discharge (Reproductive system and breast disorders) | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No